CLINICAL TRIAL: NCT04557319
Title: An Open Study of the Safety and Pharmacokinetics of GNR-038 in Sequential Dose-increase Cohorts in Healthy Volunteers
Brief Title: Safety and Pharmacokinetics of GNR-038 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CIR-HAET-I; #725 eff date 20.12.2019 (Other: Clinical trial approval number, Ministry of Health of Russia)
Record Dates: First submitted 2020-08-26; First posted 2020-09-21 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-08

CONDITIONS: Hereditary Angioedema
Keywords: Angioedema; Angioedemas, Hereditary; Vascular Diseases; Cardiovascular Diseases; Urticaria; Skin Diseases, Vascular; Skin Diseases; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases; Genetic Diseases, Inborn; Antibodies, Monoclonal; Immunologic Factors; Physiological Effects of Drugs
MeSH Terms: conditions — Angioedemas, Hereditary; Angioedema; Vascular Diseases; Cardiovascular Diseases; Urticaria; Skin Diseases, Vascular; Skin Diseases; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases; Genetic Diseases, Inborn

STUDY DESIGN:
Intervention Model Description: Sequential dose-increase cohorts in healthy volunteers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GNR-038, 25 МЕ/kg (Experimental): Recombinant C1-esterase (25 ME/kg) inhibitor intravenous infusion
  Interventions: Biological: GNR-038, 25 МЕ/kg
- GNR-038, 50 МЕ/kg (Experimental): Recombinant C1-esterase (50 ME/kg) inhibitor intravenous infusion
  Interventions: Biological: GNR-038, 50 МЕ/kg
- GNR-038, 100 МЕ/kg (Experimental): Recombinant C1-esterase (100 ME/kg) inhibitor intravenous infusion
  Interventions: Biological: GNR-038, 100 МЕ/kg

INTERVENTIONS:
Biological: GNR-038, 25 МЕ/kg — 25 МЕ/kg once per study
  Other Names: rC1inh, 25 МЕ/kg
  Arms: GNR-038, 25 МЕ/kg
Biological: GNR-038, 50 МЕ/kg — 50 МЕ/kg once per study
  Other Names: rC1inh, 50 МЕ/kg
  Arms: GNR-038, 50 МЕ/kg
Biological: GNR-038, 100 МЕ/kg — 100 МЕ/kg once per study
  Other Names: rC1inh, 100 МЕ/kg
  Arms: GNR-038, 100 МЕ/kg

SUMMARY:
It is an open-label dose-escalating study in sequential cohorts to assess safety and pharmacokinetics of GNR-038.

DETAILED DESCRIPTION:
Hereditary angioedema (HAE) is a rare potentially life-threatening genetically determined disease associated with a deficiency or impairment of C1 esterase inhibitor (C1 inhibitor) functional activity. Main clinical manifestations of HAE are recurrent mucous membranes edema and localization of the derma deep layers. Attack persist from several hours to several days and disappear without a trace in most cases, without additional therapy.

The prevalence of the disease in the world is from 1:10 000 to 1: 150 000. The plasma/recombinant C1 inhibitor use to compensate for its deficiency or insufficient functional activity in patients with HAE is recommended both for severe and for long-term and short-term (before surgical interventions and dental manipulations) prophylaxis.

GNR-038 is a recombinant C1 inhibitor (rhC1-inh), which is a complete structural and functional analogue of the plasma C1 inhibitor.

ELIGIBILITY:
Inclusion Criteria

1. Men and women aged 18 to 50 (inclusive) at the time of signing the Informed Consent Form.
2. Body mass index (BMI) in the range from 18.5 to 30 kg / m2, body weight from 50 to 90 kg.
3. The diagnosis is "healthy" according to the data of clinical and biochemical blood tests, urinalysis, results of physical examination, measurement of vital signs, results of electrocardiography.
4. Availability of written informed consent obtained from the volunteer prior to any research-related procedures performance.
5. Consent to follow the adequate contraceptive methods.

Exclusion Criteria

1. Known hypersensitivity to the components of the study drug;
2. Burdened allergic history;
3. Standard laboratory and instrumental parameters values are outside the normal range;
4. Cardiovascular, bronchopulmonary, neuroendocrine systems chronic diseases, as well as gastrointestinal tract, liver, kidneys, hematopoietic, immune systems diseases, mental illness;
5. Diseases and conditions associated with thrombosis (myocardial infarction, transient ischemic attacks, deep and superficial vein thrombosis, pulmonary embolism) less than 6 months before the screening period start, as well as an increased risk of arterial or venous thrombosis according to the investigator opinion.
6. Infection with human immunodeficiency virus (HIV), hepatitis B and C;
7. Acute infectious diseases less than 4 weeks prior to the Screening Visit;
8. Regular medication intake less than 2 weeks prior to the Screening Visit;
9. For women - the hormonal contraceptives use or hormone replacement therapy for 3 months before the screening period start;
10. Systolic pressure less than 100 mmHg or above 140 mmHg; diastolic pressure less than 70 mmHg or above 90 mmHg; pulse rate less than 60 beats/min or more than 90 beats/min;
11. Blood donation (450 ml of blood or plasma and more) less than 3 months before the Screening Visit;
12. Participation in clinical trials less than 3 months before the Screening Visit;
13. More than 10 alcohol units intake per week (1 unit of alcohol is equivalent to 1/2 liter of beer, 200 ml of wine or 50 ml of ethanol) OR anamnestic information about alcoholism, detection of ethanol in exhaled air;
14. Drug addiction, substance abuse, positive urine test for the content of potent and narcotic drugs;
15. Smoking more than 10 cigarettes a day;
16. Pregnancy or breastfeeding;
17. Other reasons that prevent the volunteer from study participating or create an unreasonable risk in the investigator opinion.

Ages: 18 Months to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | 28 Days
  Adverse events, Laboratory tests, Vital signs, Physical examination, 12-lead electrocardiogram, Allergic associated reaction, Infusion associated reaction, Antidrug antibody.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 45, 30 and 15 minutes before GNR-038 infusion; 0, 15, 30 minutes, 1, 2, 4, 8,12,16, 24, 48, 72, 96, 120,144 and 168 hours after GNR-038 infusion
  Pharmacokinetic parameters
Area under the plasma concentration versus time curve (AUC) | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8
  Pharmacokinetic parameters
Half-life (T1/2) | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8
  Pharmacokinetic parameters
Elimination rate constant (Kel) | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8
  Pharmacokinetic parameters
Mean retention time (MRT) | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8
  Pharmacokinetic parameters
Overall clearance (Cl) | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8
  Pharmacokinetic parameters
Kinetic volume of distribution (Vz) | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8
  Pharmacokinetic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Oksana A. Markova, MD, Study Chair — AO GENERIUM
Locations (1):
- State budgetary institution of healthcare of the city of Moscow "Сity polyclinic No. 2 of the Department of healthcare of the city of Moscow", Moscow, Russia

IPD SHARING:
Plan to Share IPD: No